CLINICAL TRIAL: NCT02531009
Title: A Multicenter, Prospective, Longitudinal Study to Evaluate Gastrointestinal Function and Clinical and Molecular Biomarkers in Subjects With Early and Late Diffuse Cutaneous Systemic Sclerosis, Limited Cutaneous Systemic Sclerosis, and Healthy Volunteers
Brief Title: Systemic Sclerosis Clinical and Biomarker Study
Status: Withdrawn | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 995SS001
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Healthy; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA (ribonucleic acid) will be extracted for gene expression from the skin biopsies, skin tape, and blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Approximately 10 healthy adults will be enrolled into this study
- SSc: Participants with dcSSc and lcSSc

SUMMARY:
The primary objective of the study is to assess the change in systemic sclerosis (SSc)-associated gastrointestinal (GI) tract symptoms over a 1-year period in participants with SSc.

DETAILED DESCRIPTION:
No study treatment will be administered. Study participants will continue to be treated by their respective physicians according to standard clinical practice. Data on concomitant therapy and procedures, administered as part of standard of care, will be collected at baseline and at each study visit.

ELIGIBILITY:
Key Inclusion Criteria:

Healthy volunteers

* Must be in good health as determined by the Investigator, based on medical history, physical examination, and vital signs.

Participants with diffuse cutaneous systemic sclerosis (dcSSc):

* Must fulfill the 2013 classification criteria for SSc of the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR).
* Absence of the anti-centromere autoantibody.

Participants with limited cutaneous systemic sclerosis (lcSSc):

* Must fulfill the 2013 classification criteria for SSc of the ACR and EULAR.
* Subjects with lcSSc must have disease duration of less than 5 years.

Key Exclusion Criteria:

* History of any clinically significant medical condition that can interfere with the conduct of the study, or that in the opinion of the Investigator, would compromise data interpretation.
* An active severe infection as determined by the Investigator.
* Female subjects who are pregnant or currently breastfeeding.
* A known history of malignancy.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited at participating locations in a standard clinical practice setting.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in University of California at Los Angeles Scleroderma Clinical Trial Consortium GI Tract (UCLA-SCTC GIT) instrument score in participants with SSc | Baseline to Month 12
  This participant-reported assessment is a 34-item instrument designed to measure GI tract involvement in participants with SSc. The UCLA SCTC GIT 2.0 has 7 multi-item scales: Reflux, Distension/Bloating, Diarrhea, Fecal Soilage, Constipation, Emotional Well-being, and Social Functioning and a total GIT score. All scales are scored from 0 [better health-related quality of life (HRQOL)] to 3 (worse HRQOL) except the diarrhea and constipation scales (ranges 0-2 and 0-2.5, respectively). The Total GIT Score, is developed by averaging 6 of 7 scales (excluding constipation) with lower scores indicating better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen